CLINICAL TRIAL: NCT05717595
Title: BaRiatric Surgery AnD FRUctose Handeling In Obese subjecTs
Acronym: BREADFRUIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022.0595 - NL8236601822
Record Dates: First submitted 2023-01-08; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Fructose; Glucose

STUDY DESIGN:
Intervention Model Description: randomized double blinded trial
Who Masked: Participant, Investigator
Masking Description: randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high fructose (Other): high fructose (>100 gram fructose / day) for 4 weeks
  Interventions: Dietary Supplement: fructose
- low fructose (Other): low fructose diet (<30 gram fructose intake per day isocaloric correction with dextrose) for 4 weeks
  Interventions: Dietary Supplement: fructose

INTERVENTIONS:
Dietary Supplement: fructose — oral ingestion of fructose vs dextrose
  Other Names: dextrose

SUMMARY:
To investigate whether changes in fructose dietary intake can help to improve dietary fructose-induced insulin resistance and post bariatric weight loss in obese subjects of Caucasian descent

DETAILED DESCRIPTION:
In this Randomized controlled trial, males and premenopausal women, scheduled for RYGB bariatric surgery at Spaarne Gasthuis of Caucasian Dutch descent, age ≥18 years will be put on either their high fructose diet (>100 gram fructose / day) versus a low fructose diet (<30 gram fructose intake per day isocaloric correction with dextrose) 4 weeks before bariatric surgery. For both groups, an oral (13-C labeled) fructose challenge will be performed at baseline as well as 4 weeks after start of the diet (in the week of the surgery).

Outcome measures: Primary endpoints are changes in oral fructose induced glucose and insulin postprandial plasma excursions (measured by a fructose tolerance test with 120mg 13C6-labeled fructose in relation to long term glucose handling (HOMA and Freestyle Libre) at baseline and after 4 weeks (in the week of surgery) after both diets. Secondary endpoints are changes in histology and RNA seq gene expression in liver, adipose and jejunum tissue harvested with biopsy during bariatric surgery and changes in fecal gut microbiota composition, 24h feces and urine for fructose content and (postprandial) plasma metabolites including endogenous ethanol at both timepoints. Of note, dietary intake including fructose content will be monitored by an experienced dietician from Spaarne Gasthuis. Finally, to study relations with (long term) weight loss up to 1 year after surgery related to dietary intake, the last time points at 6 and 12 months after surgery (during regular clinical outpatient visits) will be used as an exploratory endpoint to gain more insight into the relationship between gut microbiota, (pre surgery) dietary fructose intake and weight loss after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a RYGB gastric bypass*
* Men and premenopausal women > 18 years of age
* Caucasian descent
* Ability to provide written informed consent

  * All subjects on the waiting list meet the criteria for bariatric surgery, that is:
* BMI > 40 kg/m2 OR >35 kg/m2 with obesity related co-morbidity
* Reasonable supervised attempts to lose weight

Exclusion Criteria:

* Unstable metabolic condition defined as;

  * Diabetes with poor glycemic control (HbA1c > 8.5%);
  * Use of an antidiabetic or anti-obesity drug;
  * Malabsorptive or restrictive bariatric (weight loss) surgery in history
* Evidence for a form of liver disease (except for NAFLD without cirrhosis)
* Known genetic basis for insulin resistance or glucose intolerance
* Use of certain drugs known to produce hepatic steatosis in the previous 6 months (such as oral corticosteroids, high-dose estrogens, methotrexate, tetracycline, amiodarone)
* Malabsorptive disease orders (celiac disease, inflammatory bowel disease)
* Use of certain drugs that may injure the lining of the intestine in the previous months (colchicine, cholestyramine)
* Excessive alcohol intake (≥5 IU per day or ≥ 14 IU per week)
* Recent use of antibiotics (≤ 3 months before surgery)
* Hemostasis disorders or current treatment with anticoagulants Any primary lipid disorder
* Unable to maintain diet intervention, or unable to reliably rapport diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
oral fructose handling | 4 weeks
  to correlate changes in oral fructose excursions (measured by AUC of fructose tolerance test enriched with 13C6-labeled fructose with glucose excursions (MAGE by Freestyle Libre)

SECONDARY OUTCOMES:
fructose changes in visceral organs | 4 weeks up to one year
  to correlate with changes in histology and RNA seq gene expression in liver, adipose and jejunum tissue harvested with biopsy during bariatric surgery
gutmicrobiota | 4 weeks up to one year
  to correlate with changes in fecal gut microbiota composition
metabolites | 4 weeks up to one year
  to correlate with (postprandial) plasma metabolites including endogenous ethanol
weight | 4 weeks up to one year
  to correlate with with (long term) weight loss at 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
not allowed due to GDPR in Netherlands